CLINICAL TRIAL: NCT05867433
Title: Strong Teens for Healthy Schools Change Club: A Civic Engagement Approach to Improving Physical Activity and Healthy Eating Environments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB2022-1159D; R01MD018214 (NIH)
Record Dates: First submitted 2023-04-11; First posted 2023-05-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Diseases; Nutrition; Physical Activity
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: School-based cluster randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STHS Intervention (Experimental): Participants in this group (10 schools) will participate in the STHS program.
  Interventions: Behavioral: STHS Intervention
- Usual Care (Other): Participants in this group (10 schools) will continue with usual care, as they will not be asked to add or remove any of their current, physical activity, healthy eating, or positive youth development programming.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: STHS Intervention — STHS program
  The intervention group (10 schools) will participate in the STHS program. During the fall semester (September to December), the intervention group will receive 24 thirty-minute modules (or twelve 1-hour modules) that provide education on civic engagement, healthy eating, and physical activity. During the spring semester (February to May), the intervention group will receive 24 thirty-minute modules (or twelve 1-hour modules) that focus on implementing the school health environmental change project and receive support for maintaining individual-level healthy eating and physical activity behaviors.
  Arms: STHS Intervention
Behavioral: Usual Care — No STHS program
  The usual care group will be offered the same activities as the intervention group after the conclusion of the research study.
  Arms: Usual Care

SUMMARY:
Strong Teens for Healthy Schools (STHS) is a school-based, civic engagement program that empowers middle school students to improve their physical activity and healthy eating behaviors, improve their cardiovascular disease outcomes, and create positive change in their school health environments.

DETAILED DESCRIPTION:
The investigators will conduct a cluster-randomized controlled trial to evaluate the impact of the Strong Teens for Healthy Schools (STHS) program on cardiovascular disease-related outcomes. STHS is a multi-level, theory-based civic engagement program to catalyze positive food and physical activity environmental change and improve cardiovascular disease-related health (CVD) outcomes among 6th and 7th-grade students.

Title 1 middle schools in Texas (n=20) with > 40% Hispanic and Black students will be randomized at baseline to the intervention condition (STHS program) or control condition (will continue with usual care, as they will not be asked to add or remove any of their current, physical activity, healthy eating, or positive youth development programming) (n=20-25 students per school).

The investigators hypothesize that students who participate in STHS will have reduced MetS risk, improved positive youth developmental outcomes, and improved social and environmental outcomes immediately post-intervention and one year after study completion compared to students in a control condition.

ELIGIBILITY:
School Inclusion Criteria:

* > 50 6th and 7th grade students
* > 40% economically disadvantaged students
* > 40% Black and Hispanic students

School Exclusion Criteria:

Student Inclusion Criteria:

* 6th or 7th grade student
* Attend a Title 1 middle school that is participating in the STHS intervention
* Read and understand English

Student Exclusion Criteria:

* Participation in a weight loss program in the past 3 months
* Presence of a condition that prevents participation in physical activity

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of metabolic syndrome (MetS) | Baseline, 9 months (immediate post intervention), 4 months and 12 months post intervention
  MetS is present after identifying abdominal obesity plus at least two of the four other MetS Risk factors: high blood pressure, high blood sugar, low HDL cholesterol, and high triglyceride levels.
  MetS = (abdominal obesity) + (2 of 4 other MetS Risk factors)
  Measures to determine MetS risk factors:
  1. Abdominal obesity: waist circumference >90th percentile for child's sex and age
  2. High blood pressure: systolic blood pressure ≥130 mm Hg or diastolic blood pressure ≥90 mmHg)
  3. High blood glucose: blood glucose ≥5.6 mmol/L or known diabetes
  4. Low HDL cholesterol: HDL cholesterol <1.03 mmol/L
  5. High triglyceride level: Triglyceride level ≥ 1.7mmol/L
Change in the number of MetS risk factors | Baseline, 9 months (immediate post intervention), 4 months and 12 months post intervention
  Change in the number of MetS risk factors = (new # of MetS risk factors) - (original # of MetS risk factors)
  Measures to determine MetS risk factors:
  1. Abdominal obesity: waist circumference >90th percentile for child's sex and age
  2. High blood pressure: systolic blood pressure ≥130 mm Hg or diastolic blood pressure ≥90 mmHg)
  3. High blood glucose: blood glucose ≥5.6 mmol/L or known diabetes
  4. Low HDL cholesterol: HDL cholesterol <1.03 mmol/L
  5. High triglyceride level: Triglyceride level ≥ 1.7mmol/L
Positive Youth Development score | Baseline, 9 months (immediate post intervention), 4 months and 12 months post intervention
  Positive youth development will be measured using a 5 C's Model of Positive Youth Development Scale-Short Form (PYD-SF): A 34-item scale that assesses the strength of psychological, behavioral, and social development in youth.
  The five dimensions measured are:
  1. Competence (sense of proficiency)
  2. Confidence (self-worth, self-efficacy)
  3. Character (adherence to societal and cultural rules)
  4. Connection (bonds with people and institutions)
  5. Caring (sympathy and empathy towards others)

SECONDARY OUTCOMES:
Blood pressure level | Baseline, 9 months (immediate post intervention), 4 months and 12 months post intervention
  Blood pressure (systolic and diastolic) will be measured with two numbers using an automated Omron sphygmomanometer.
Concentration of blood glucose | Baseline, 9 months (immediate post intervention), 4 months and 12 months post intervention
  Glucose will be measured using a portable Cholestech LDX analyzer to assess a single capillary blood sample following an overnight fast.
Waist circumference | Baseline, 9 months (immediate post intervention), 4 months and 12 months post intervention
  Waist circumference will be measured at the midpoint between the floating rib and iliac crest using a tape measure.
Concentration of HDL cholesterol | Baseline, 9 months (immediate post intervention), 4 months and 12 months post intervention
  HDL-C will be measured using a portable Cholestech LDX analyzer to assess a single capillary blood sample following an overnight fast.
Concentration of serum triglycerides | Baseline, 9 months (immediate post intervention), 4 months and 12 months post intervention
  Triglycerides will be measured using a portable Cholestech LDX analyzer to assess a single capillary blood sample following an overnight fast.
Height | Baseline, 9 months (immediate post intervention), 4 months and 12 months post intervention
  Height will be measured using a stadiometer in inches.
Weight | Baseline, 9 months (immediate post intervention), 4 months and 12 months post intervention
  Weight will be measured with a scale in pounds.
Body mass index (BMI) | Baseline, 9 months (immediate post intervention), 4 months and 12 months post intervention
  Weight will be measured with a scale, and height will be measured using a stadiometer. BMI will be calculated as BMI = (weight (lb)/height (inches)2) x 703.
Concentration of subdermal carotenoids | Baseline, 9 months (immediate post intervention), 4 months and 12 months post intervention
  The concentration of subdermal carotenoids will assess the changes in fruit and vegetable consumption using the Veggie Meter: A non-invasive, portable machine that measures subdermal carotenoid levels using resonance Raman spectroscopy.
Accelerometer-derived physical activity estimation | Baseline to 9 months
  Physical activity will be measured using Actigraph accelerometers. Measurements will include light physical activity (PA), moderate PA, moderate to vigorous PA, and vigorous PA.
Sedentary time | Baseline to 9 months
  Sedentary time will be measured using Actigraph accelerometers.
Time spent sleeping | Baseline to 9 months
  Sleep time will be measured using Actigraph accelerometers.
Physical fitness capacity estimation | Baseline, 9 months (immediate post intervention), 4 months and 12 months post intervention
  Physical fitness will be measured using the FitnessGram PACER multistage aerobic capacity test: Children will run back and forth 20 meters, with an initial running speed of 8.5 km/hour and a progressive 0.5-km/hour increase in running speed every minute. As the test continues it becomes progressively harder. The number of laps completed is used to estimate children's physical fitness physical fitness.
School physical activity and nutrition environment assessment | Baseline to 9 months
  The school's physical activity and nutrition environments will be measured using a self-reported School Environment Survey.
Assessment of perceptions of school environments and school-specific dietary intake patterns | Baseline to 9 months
  Perceptions related to physical activity and nutrition within the school setting will be measured using the Perceptions of the Environment and Patterns of Diet at School (PEA-PODS) survey.
Assessment of perceived sociopolitical control | Baseline to 9 months
  Perceived sociopolitical control will be measured using the Youth Engagement and Action for Health (YEAH!) survey. The YEAH survey will be used to assess students' perceived sociopolitical control (i.e., participation in advocacy programs and optimism for change).
Assessment of assertiveness | Baseline to 9 months
  Assertiveness will be measured using the Youth Engagement and Action for Health (YEAH!) survey. The YEAH survey will be used to assess students' assertiveness (i.e., ability to engage with adults and peers).
Assessment of participatory competence and decision-making | Baseline to 9 months
  Participatory competence and decision-making will be measured using the Youth Engagement and Action for Health (YEAH!) survey. The YEAH survey will be used to assess students' participatory competence and decision-making (i.e., ability to influence group decision-making).
Assessment of advocacy outcome efficacy | Baseline to 9 months
  Advocacy outcome efficacy will be measured using the Youth Engagement and Action for Health (YEAH!) survey. The YEAH survey will be used to assess students' advocacy outcome efficacy (i.e., belief in their ability to work with others to improve the school's physical activity and nutrition environment).
Peer concentration of subdermal carotenoids | Baseline to 9 months
  The concentration of subdermal carotenoids will assess peers' engagement in health behaviors changes in fruit and vegetable consumption using the Veggie Meter: A non-invasive, portable machine that measures subdermal carotenoid levels using resonance Raman spectroscopy.
Peer Body mass index (BMI) | Baseline to 9 months
  Peers' engagement in health behaviors will be measured by the change in peers' BMI. Weight will be measured with a scale, and height will be measured using a stadiometer. Calculate BMI with the formula: BMI = (weight (lb)/height (inches)2) x 703.
Peer physical fitness capacity estimation | Baseline to 9 months
  Peers' engagement in health behaviors will be measured by the change in peers' physical fitness. Physical fitness will be measured using the FitnessGram PACER multistage aerobic capacity test: Children will run back and forth 20 meters, with an initial running speed of 8.5 km/hour and a progressive 0.5-km/hour increase in running speed every minute. As the test continues it becomes progressively harder. The number of laps completed is used to estimate children's physical fitness physical fitness.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M AgriLife Dallas Center, Dallas, Texas, United States

REFERENCES:
- [Derived] MacMillan Uribe AL, George A, McNeely A, Xin L, Largacha Cevallos E, Rethorst C, Seguin Fowler RA, Szeszulski J. Strong Teens for Healthy Schools: Protocol for evaluating a youth nutrition, physical activity, and civic engagement protocol. Front Public Health. 2025 Sep 17;13:1654678. doi: 10.3389/fpubh.2025.1654678. eCollection 2025. PMID 41041380